CLINICAL TRIAL: NCT02445014
Title: Pilot Study for Imaging of Barrett's Esophagus Using an Spectrally Encoded Confocal Microscopy Tethered Endoscopic Capsule
Brief Title: Pilot Study to Image the Esophagus Using a SECM Tethered Endoscopic Capsule
Acronym: SECM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2014-P-002058; 1R01CA184102-01 (NIH)
Record Dates: First submitted 2015-04-16; First posted 2015-05-15 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Healthy; Barrett's Esophagus; Gastric Acid Reflux
Keywords: Barrett's; GERD; Capsule; SECM
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MGH SECM Imaging Capsule (Experimental): Subject will swallow the SECM imaging capsule and images will be acquired using the SECM Imaging system.
  Interventions: Device: MGH SECM Imaging Capsule

INTERVENTIONS:
Device: MGH SECM Imaging Capsule — Imaging of the Esophagus using the SECM capsule and SECM Imaging system

SUMMARY:
The goal of this research is to test the imaging quality of the modified, larger diameter, tethered Spectrally Encoded Confocal Microscopy (SECM) capsule in healthy subjects, subjects with Barrett's Esophagus (BE), and subjects with Gastroesophageal reflux disease (GERD).

DETAILED DESCRIPTION:
36 subjects including 12 healthy volunteers, 12 patients with Barrett's Esophagus and 12 with Gastroesophageal reflux disease will be enrolled and asked to swallow the SECM HITEC Capsule. The subjects will be awake and unsedated.

The capsule is attached to a string like tether which allows the operator to control as well as navigate the capsule as it progresses down the esophagus using natural propulsive force called peristalsis.

As the capsule progresses through the esophagus, multiple images of the esophagus are acquired in real time to be analyzed later.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 1) a healthy volunteer (18 years or older), or 2) a subject with prior diagnosis of BE (18 years or older), or 3) a subject with prior diagnosis of GERD (18 years or older).
* AND Subject must be able to give informed consent.
* AND Subject must eat no solid foods for 8 hours before the procedure and only clear liquids for 2 hours before the procedure.

Exclusion Criteria:

* Subjects with any history of or known upper gastrointestinal strictures
* OR Subjects with a history of Crohn's disease,
* OR Subjects with difficulty swallow

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD., PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study we were trying to establish how many participants can provide us with quality imaging using this new technology. Therefore we treated them as one group. 2 healthy subjects and one with BE were enrolled.
  Upon reviewing imaging data it was concluded that this new technology is not optimal for the study and the enrollment was stopped.
Period: Overall Study
Arm/Group | MGH SECM Imaging Capsule
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- MGH SECM Imaging Capsule: Subject will swallow the new large SECM imaging capsule and images will be acquired using the SECM Imaging system.
Arm/Group | MGH SECM Imaging Capsule
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility for Imaging of Esophagus Using an SECM Tethered Endoscopic Capsule.
Description: The number of subjects from whom successful SECM imaging was obtained
Time Frame: 20 minute visit (5-7 minute imaging)
Measure: Count of Participants; unit: Participants
Arm/Group | MGH SECM Imaging Capsule
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: During the procedure and 10 minutes after
Groups:
- MGH SECM Imaging Capsule: Subject will swallow the SECM imaging capsule and images will be acquired using the SECM Imaging system. The imaging quality will be reviewed.
Arm/Group | MGH SECM Imaging Capsule
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No